CLINICAL TRIAL: NCT02486679
Title: Cervical Ripening at Term With Prostaglandin E2 Tablets Versus Foley Catheter: a Randomized Controlled Trial
Brief Title: A Trial of Prostaglandin E2 Tablets Versus Foley Catheter for Labor Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wolfson Medical Center (Other Government)
Responsible Party: Principal Investigator, Hadas Ganer Herman, MD, Wolfson Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0095-15-WOMC
Record Dates: First submitted 2015-06-22; First posted 2015-07-01 (Estimated); Last update posted 2016-04-29 (Estimated); Status verified 2016-04

CONDITIONS: Labor, Induced
MeSH Terms: interventions — KLK15 protein, human; Dinoprostone; Tablets

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PGE2 (Active Comparator): Patients allocated to vaginal PGE2 (Prostin) for cervical ripening
  Interventions: Drug: Prostin (PGE2) tablets
- Foley catheter (Active Comparator): Patients allocated to foley catheter placement for cervical ripening
  Interventions: Device: Foley catheter

INTERVENTIONS:
Drug: Prostin (PGE2) tablets
  Arms: PGE2
Device: Foley catheter
  Arms: Foley catheter

SUMMARY:
A randomized controlled trial comparing labor induction with vaginal PGE2 tablets and foley catheter for cervical ripening.

ELIGIBILITY:
Inclusion Criteria:

* Singleton term pregnancies (>37 weeks), vertex presentation
* Intact membranes
* Low Bishop score (<7)
* First, second or third delivery
* Medical indication for induction
* Viable fetus

Exclusion Criteria:

* Contraindication for vaginal delivery, for PGE2 or foley catheter
* Gestational age<37 weeks, premature rupture of membranes, fetal or uterine malformations, previous cesarean section, uncertain dating, unwilling to participate in trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-07 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Time to active labor | Post labor- up to 24 hours
  Hours from foley cather placement or first PGE2 tablet placment to active labor, defined as cervical dilitation >4 cm and/or cervical effacement>80%

SECONDARY OUTCOMES:
Delivery within 24 hours | post-labor - up to 24 hours
  Delivery within 24 hours from foley catheter /first PGE2 tablet palcement
Cesarean section rate | post labor - up to 24 hours
  Delivery via cesarean section
Maternal complications | participants will be followed for labor course and the duration of hospital stay, an expected average of 5 days
  Documented complications during labor, including: excessive hemmorhage, infection (chorioamnionitis)
Neonatal complications | Neonates of participants will be followed for labor course and the duration of hospital stay, up to 1 month
  Documented complications such as non-reassuring fetal heart rate, fetal pH, NICU admission, early neonatal sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Edith Wolfson Medical Center, Holon, Israel